CLINICAL TRIAL: NCT01913106
Title: Phase I-II Study HSV-tk + Valacyclovir Therapy in Combination With Brachytherapy for Recurrent Prostate Cancer With or Without Metastatic Disease
Brief Title: HSV-tk + Valacyclovir Therapy in Combination With Brachytherapy for Recurrent Prostate Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00000601; IRB 0107-0009 (Other: Houston Methodist Research Institute IRB)
Record Dates: First submitted 2013-07-25; First posted 2013-07-31 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HSV-tk + Valacyclovir and Brachytherapy (Experimental): You will be given an antibiotic (Ciproflaxin) to take twice a day beginning the day before the procedure, and continuing for a total of 3 - 5 days. You will also be given 4 pills called (Valtrex) valacyclovir to take three times a day for 14 days, beginning the day before the procedure. You will be given a pill diary in which you will record each dose of valacyclovir that you take. You will receive brachytherapy (radioactive seed placement) the day after you begin taking your pills. After the radioactive seeds are placed, while you are still in the operating room, you will receive an injection into your prostate of 1 or 2 ml (one-fifth or two-fifths of a teaspoon) of a solution of the vector carrying the gene.
  Interventions: Drug: HSV-tk +Valacyclovir in Combination with Brachytherapy

INTERVENTIONS:
Drug: HSV-tk +Valacyclovir in Combination with Brachytherapy — The investigators insert a gene from a herpes simplex virus (HSV), which is a small piece of the basic structure of the virus, into the prostate gland tumor cells. The gene is called the thymidine kinase (tk) gene, which the cell uses to make a protein that can change valacyclovir, The way the tk gene will be transported into the tumor cells is by using a vector or "vehicle" to carry the tk gene into the cells. In this case the vector is a virus - an adenovirus. Scientists at the Department of Cell and Gene Therapy at The Methodist Hospital removed a portion of the adenovirus' genetic material that allows it to replicate so that it cannot cause infections. In place of the removed genetic material the scientists inserted the tk gene. Now the vector can carry the tk gene into tumor cells. When the vector/gene combination gets into tumor cells, it inserts itself into the cells' command center (nucleus) and tells the tumor cells to begin making thymidine kinase protein.
  Other Names: IND 13567

SUMMARY:
The purpose of this study is to conduct a Phase I - II clinical trial to extend preclinical studies involving in situ HSV-tk + Valacyclovir gene therapy in combination with brachytherapy for recurrent prostate cancer. This will provide a novel therapeutic approach to prostate cancer and hopefully impact on the development of metastatic disease and the control of preexisting metastasis.

DETAILED DESCRIPTION:
This investigational new drug application describes a proposed phase I/II study designed to assess the safety and efficacy of AdV-tk gene therapy in combination with standard brachytherapy for patients with locally recurrent prostate cancer after having failed radiation as a primary treatment with or without minimal metastasis. These patients do not have any standard treatment that has been demonstrated to have a high degree of efficacy in eradicating the tumor with a reasonable degree of safety. Thus, the potential risks associated with the use of gene therapy in this group would appear reasonable. This application is for use of a replication defective adenovirus vector (ADV/RSV-tk) delivering the HSV-tk gene as a biologic vector for gene therapy.

Direct introduction of therapeutic genes into malignant cells in vivo may provide an effective treatment of solid tumors such as prostate cancer. The herpes simplex virus thymidine kinase (HSV-tk) gene codes for an enzyme which phosphorylates the nucleoside analog ganciclovir (GCV) into an intermediate that is incorporated into newly synthesized DNA and terminates further replication, leading to cell death. Since normal mammalian cells do not possess this enzyme, cytotoxicity depends on the successful introduction and expression of the HSV-tk gene, phosphorylation of ganciclovir and synthesis of DNA. Non-dividing cells may express HSV-tk and phosphorylate ganciclovir but are not harmed since they do not synthesize DNA. This approach is especially suitable for the treatment of tumors where rapidly dividing tumor cells are adjacent to tissues made up largely of non-proliferating cells. Using human and animal models for prostate cancer we have demonstrated that adenovirus-mediated transfer of the HSV-tk gene resulted in sensitivity to ganciclovir in vitro and growth suppression of mouse prostate cancer in vivo.

ELIGIBILITY:
INCLUSION CRITERIA:

* biopsy-proven local recurrence of prostate cancer without metastatic disease after the hormone therapy at least 2 year after the completion of definitive radiation therapy
* Zubrod performance status 0-1
* WBC ≥ 4,000/μl, platelets ≥ 100,000/μl
* hemoglobin ≥ 8.5 mg/dl
* normal partial thromboplastin time and prothrombin time
* bilirubin < 1.5 mg/dl, and AST and alanine aminotransferase < 2.5 times the upper limit of normal
* Serum creatinine ≤ 1.6 mg/dl
* Must undergo pre-treatment evaluation of tumor extent and tumor measurement
* Nutritional and general physical condition must be considered compatible with the proposed radio-therapeutic treatment
* Not on any other experimental therapeutic cancer treatment
* No active untreated infection
* No major medical or psychiatric illness
* International Prostate Symptom Score (IPSS) less than 15
* Signed study-specific consent form prior to study entry
* Prostate volume less than 50 cc
* PSA > 10ng/ml within the past 3 months may enter study

EXCLUSION CRITERIA:

* Symptomatic metastasis disease
* Patients with a life expectancy < 10 years
* Patients on corticosteroids or any immunosuppressive drugs.
* HIV + patients
* Patients with acute infections (viral, bacterial, or fungal infections requiring therapy)
* Patients with cirrhosis.
* Patients with collagen vascular diseases
* International Prostate Symptom Score (IPSS) greater than 15
* Prostate volume greater than 50 cc
* Second active cancer except cutaneous cancer
* Patients with history of allergies to valacyclovir, acyclovier or who cannot take oral pills

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2007-06; Primary Completion 2018-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
1. Safety based on standard laboratory and clinical adverse event monitoring | 5-year biochemical disease free survival rate

SECONDARY OUTCOMES:
Local control survival (measured by PSA and biopsy) | 5-year biochemical disease free survival rate
Evaluate immunological markers | 5-year post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Edward B Butler, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No